CLINICAL TRIAL: NCT03358446
Title: The Optimal Leg Angulation of Femoral Central Catheterization in Pediatrics
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-09-027
Record Dates: First submitted 2017-11-26; First posted 2017-11-30 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2017-09

CONDITIONS: Pediatric Disorder; Femoral Artery Injury; Emergencies
Keywords: central catheterization; femoral vein central catheterization; leg angulation
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A group: Based on the presence of non-overlapping range between femoral artery and vein from the initial observation, the patients were divided into following two groups.
  A group is the patients with non-overlapping range
  Interventions: Other: A group
- S group: S group is the patients without non-overlapping range
  Interventions: Other: S group

INTERVENTIONS:
Other: A group — The optimal range of leg abduction was defined as the range without overlap in A group and the range presenting that the overlap was less-than half of the diameter of femoral vein in S group.
  A1 angle defined the point that the femoral vein and artery started non-overlapping interval when increasing the angle of the leg in the A group and the A2 angle is defined the point that the femoral vein and artery ended non-overlapping interval.
  Groups: A group
Other: S group — B1 is the angle at which the overlap starts at the half of the femoral vein radius when increasing the angle of the leg in the S group, B2 is the angle at which overlap starts at half or more of the femoral vein radius again. In the range of B1 and B2 angles, they are overlapped by half or less of the femoral vein radius.
  Groups: S group

SUMMARY:
Evaluation for the range of smallest leg angulation with femoral artery and vein overlap with femoral central catheterization in pediatrics.

DETAILED DESCRIPTION:
In pediatrics, femoral vein catheterization often overlaps with the femoral artery.

In this case, the risk of artery puncture is high, vein collapse when artery puncture 2nd, 3rd times exceeds the success rate of catheterization becomes low. In previous study, comparing 0, 30, and 60 degrees with frog leg position, there was a study that the overlap was the smallest at 60 degrees. A previous study was a simple frog leg position and a study in fragmented predetermined angles. On a continuous measurement, we planned the study under the assumption that there is a more definite range of optimal angulation.

Ultrasound probe in the state of Inguinal crease, we find a part without bifurcation of femoral artery and femoral vein in frog leg position(external rotation + flexion increase). Increase the leg angle and check the vein and arterie relations.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients younger than 3 years
2. ASA class 1-3
3. Patients scheduled for elective surgery.
4. If the patient's guardian can understand and write the contents of the agreement.

Exclusion Criteria:

1. A patient with previous history of dislocation of the hip.
2. Hip joints with limited hip movement.
3. A patient with vascular malformation of the femoral vein
4. Emergency surgery
5. Hemodynamic unstable patient
6. If the patient's guardian cannot understand and write the contents of the agreement.

Max Age: 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients scheduled for elective surgery.
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
A range of angles in which arteries and veins do not overlap | Intraoperative ( after anesthesia induction)
  The optimal range of leg abduction was defined as the range without overlap in A group and the range presenting that the overlap was less-than half of the diameter of femoral vein in S group.

CONTACTS AND LOCATIONS:
Overall Officials: jonghwan lee, MD, PhD, Principal Investigator — Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Samsung Medical Center, Sungkyunkwan University, School of Medicine, Seoul, South Korea